CLINICAL TRIAL: NCT02079428
Title: The National Registry Study of Hospitalized Heart Failure Patients in China
Brief Title: China National Heart Failure Registry
Acronym: CN-HF
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shanghai Institute of Cardiovascular Diseases (Other)
Responsible Party: Sponsor
Other Study IDs: 2011BAI11B10
Record Dates: First submitted 2014-03-02; First posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-03

CONDITIONS: Cardiac Failure; Congestive Heart Failure
Keywords: Heart Failure; Registry; China
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Systolic heart failure, Diastolic heart failure
  Interventions: Other: No interventions

INTERVENTIONS:
Other: No interventions

SUMMARY:
The purpose of CN-HF is to establish the national registration of hospitalized heart failure patients, evaluate and compare the clinical features and prognosis of diastolic and systolic heart failure, and find out the status of treatment and implementation of guidelines on heart failure in China.

DETAILED DESCRIPTION:
The CN-HF is a national, multi-centered, prospective and observational registry study, led by Shanghai Institute of Cardiovascular Diseases, Zhongshan Hospital (head unit) with 50 to 100 secondary and tertiary hospitals involved. The study planed to consecutively enroll 10 000 heart failure patients fulfilling the inclusion criteria. Each center will register all patients with heart failure involved in the discharge or death diagnosis in consecutive 6 months, and each registered patient will be followed up for at least 3 years. The study consists 3 phases: the screening phase, the baseline registry phase, and the follow-up registry phase.

The data collecting and reporting will employ the combination of paper-based case report form (CRF) and web-based electronic CRF. The handwriting paper CRF are provided by the head unit as raw data. Investigators in each center should input the raw data into the web-based CRF using the login name and password provided by the head unit.

The data management center specified by the head unit is responsible for the establishment and maintenance of CRF and the central database, the regular check of data submitted and the updating of the database. During the data collection, the data management center will also regularly check and report errors in the CRF and feedback to each centers and supervise to correct errors.

At the end of the study, the database will be locked after all data being checked and updated. Each participating center will preserve their own copy of paper-based CRF and electronic CRF, the head unit will preserve all paper-based CRFs and electronic CRFs.

Statistical analysis will be performed by independent statisticians in the head unit (Shanghai Institute of Cardiovascular Diseases) using the SAS software. The Student t test or chi-square test will be used for comparison between two groups. The Cox proportional hazard model will be used to investigate the risk factors for adverse cardiovascular events.

ELIGIBILITY:
Inclusion Criteria:

* Patients discharged from the department of cardiology;
* Discharge or death diagnosis involves diseases with I50 as the beginning of the International Classification of Diseases (ICD)-10 code, including congestive heart failure, congestive heart disease, cardiac failure, right side heart failure, right side ventricular failure, acute left side heart failure, chronic left side cardiac dysfunction, cardiac asthma, left side heart failure, left side heart failure with acute pulmonary edema, low cardiac output syndrome, cardiac dysfunction, acute heart failure, chronic heart failure, grade Ⅱ cardiac function class, grade Ⅲ cardiac function class, grade Ⅱ-Ⅲ cardiac function class, grade Ⅳ cardiac function class, heart failure, cardiac-renal failure, circulatory failure, and grade Ⅰcardiac function class (I51.903), pregnancy with heart failure (O99.408), pregnancy with cardiac dysfunction (O99.429), postpartum cardiac dysfunction (O99.434), post-operative heart failure with pulmonary edema (I97.104), and heart failure after cardiac surgery (I97.106);
* Agree to sign an informed consent form.

Exclusion Criteria:

* Refuse to sign an informed consent form;
* Already involved in this study during previous hospitalization.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study planed to consecutively enroll 10 000 heart failure patients fulfilling the inclusion criteria. Each center will register all patients with heart failure involved in the discharge or death diagnosis in consecutive 6 months.
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2013-01; Primary Completion 2016-06 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Number of death | 36 months after index discharge

SECONDARY OUTCOMES:
Number of patients rehospitalized for worsened heart failure | 36 months after index discharge

OTHER OUTCOMES:
Change from baseline in New York Heart Association (NYHA) cardiac function classes | 36 months after index discharge

CONTACTS AND LOCATIONS:
Overall Officials: Jingmin Zhou, Professor, Principal Investigator — Shanghai Institute of Cardiovascular Diseases, Zhongshan Hospital, Fudan University
Locations (1):
- Shanghai Institute of Cardiovascular Diseases, Zhongshan Hospital, Fudan University, Shanghai, China

REFERENCES:
- [Derived] Zhou J, Cao J, Jin X, Zhou J, Chen Z, Xu D, Yang X, Dong W, Li L, Fan Y, Chen L, Zhong Q, Fu M, Hu K, Ge J; CN-HF investigators. Digoxin is associated with worse outcomes in patients with heart failure with reduced ejection fraction. ESC Heart Fail. 2020 Feb;7(1):138-146. doi: 10.1002/ehf2.12539. Epub 2020 Jan 29. PMID 31994361
- [Derived] Jin X, Cao J, Zhou J, Wang Y, Han X, Song Y, Fan Y, Chen Z, Xu D, Yang X, Dong W, Li L, Chen L, Zhong Q, Fu M, Hu K, Zhou J, Ge J; CN-HF investigators. Outcomes of patients with anemia and renal dysfunction in hospitalized heart failure with preserved ejection fraction (from the CN-HF registry). Int J Cardiol Heart Vasc. 2019 Aug 31;25:100415. doi: 10.1016/j.ijcha.2019.100415. eCollection 2019 Dec. PMID 31508483